CLINICAL TRIAL: NCT00790309
Title: Hormonal and Inflammatory Parameters Affecting Early Diabetes Resolution Following Weight Loss Surgery
Brief Title: Early Diabetes Resolution After Weight Loss Surgery
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Naji Abumrad, Chairman, Department of Surgery, Vanderbilt University Medical Center
Other Study IDs: NNA-Early DM Resolution
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Diabetes
Keywords: Obesity; Diabetes; Bariatric surgery
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Weight loss surgery: This group will be comprised of people having weight loss surgery: Roux-en Y gastric bypass, vertical sleeve gastrectomy, or adjustable gastric banding
  Interventions: Procedure: Weight loss surgery
- Abdominal surgery: This group will be comprised of people having abdominal surgeries such as nissen fundoplication or cholecystectomy.
  Interventions: Procedure: Laparoscopic abdominal surgeries
- Lean: This group will be comprised of normal weight healthy volunteers.

INTERVENTIONS:
Procedure: Weight loss surgery — Weight loss surgery
  Groups: Weight loss surgery
Procedure: Laparoscopic abdominal surgeries — laparoscopic abdominal surgeries
  Groups: Abdominal surgery

SUMMARY:
The primary objective is to compare inflammatory, hormonal, and metabolic changes in the very short term after various bariatric surgical procedures (Roux-en Y Gastric Bypass, Vertical Sleeve Gastrectomy, and Adjustable Gastric Banding)and other abdominal surgeries, as well as to compare these changes to diet-induced changes in the same population.

ELIGIBILITY:
Inclusion Criteria for surgery groups:

* BMI of 30 kg/m2 or higher
* Ages 18-65
* History of impaired glucose tolerance or T2DM

Inclusion Criteria for normal weight group:

* BMI of 30 kg/m2 or lower
* Ages 18-65

Exclusion Criteria:

* Development of an intercurrent infection
* Prior gastric, duodenal, proximal jejunal surgery or pancreas resection
* Current use of thiazolidinediones
* Current use of dipeptidyl peptidase-IV inhibitors (e.g., sitagliptin) or glucagon-like peptide-1 analogs (e.g., exenatide)
* Any condition felt by the PI or co-investigators to interfere with ability to complete the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects scheduled for weight loss surgery or other abdominal surgeries will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2008-12; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Determine to what extent improvements in glycemic control can be attributed to caloric restriction after weight loss surgery | 10 days post-op

SECONDARY OUTCOMES:
Determine changes in inflammatory markers after weight loss surgery | 10 days post-op

CONTACTS AND LOCATIONS:
Overall Officials: Naji Abumrad, MD, Principal Investigator — Vanderbilt University Medical Center

REFERENCES:
- [Derived] Garcia AE, Kasim N, Tamboli RA, Gonzalez RS, Antoun J, Eckert EA, Marks-Shulman PA, Dunn J, Wattacheril J, Wallen T, Abumrad NN, Flynn CR. Lipoprotein Profiles in Class III Obese Caucasian and African American Women with Nonalcoholic Fatty Liver Disease. PLoS One. 2015 Nov 23;10(11):e0142676. doi: 10.1371/journal.pone.0142676. eCollection 2015. PMID 26599819